CLINICAL TRIAL: NCT06753604
Title: Investigation of the Relationship Between Gremlin-1 Levels and Wagner Classification inDiabetic Foot Patients and Evaluation of Its Usability as a Biomarker in the Progress toAmputation
Brief Title: Gremlin-1 and Wagner Classification: Potential Biomarker for Amputation in Diabetic Foot Patients
Status: Completed | Type: Observational
Sponsor: Seyma Acik (Other)
Collaborators: Ege University (Other)
Responsible Party: Sponsor-Investigator, Seyma Acik, Principal Investigator Medical Doctor, Ege University
Organization: Ege University (Other)
Other Study IDs: TTU-2020-21555
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus; Diabetic Foot Disease; Diabetic Foot Ulcer; Diabetic Neuropathy; Peripheral Arterial Disease
Keywords: diabetic foot; gremlin-1; amputation
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetic Neuropathies; Peripheral Arterial Disease; Polyposis Syndrome, Hereditary Mixed, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with diabetic foot: Patients were divided into groups according to the stage of diabetic foot ulcer. Patients were staged according to the Wagner classification.

SUMMARY:
The aim of the approach to diabetic foot patients is to heal the wound, mobilize the patient, increase the quality of life, and reduce DA-related amputations as much as possible. For this purpose, early diagnosis and early intervention with multidisciplinary treatment methods are important. There is no marker used to determine the prognosis, predict the progression to amputation, and take precautions for diabetic foot.

Based on this need, investigators planned to examine the gremlin-1 level in patients with diabetic foot wounds by grouping them according to the severity of the disease (according to the Wagner classification). There is no previous study examining the relationship between gremlin-1, which has been shown to play a role in inflammation, fibrosis, and angiogenesis, and diabetic foot.

In this study, investigators aimed to show the relationship between gremlin-1 in diabetic foot and Wagner classification and its usability as a biomarker in progression to amputation. Being the first study to be conducted on this subject in the literature increases the importance of the project.

DETAILED DESCRIPTION:
Diabetic foot (DA), a microvascular complication of diabetes mellitus (DM), is a significant cause of morbidity and mortality. While the prevalence of diabetic foot is reported to be between 4 and 10%, the lifetime risk of developing DA in a person diagnosed with diabetes is as high as 25%. Diabetic foot wounds lead to deterioration of the patient's quality of life, loss of work power, psychosocial trauma, and increased health care costs. These are the most common causes of hospitalization and longest hospital stay in diabetic patients. 50-70% of non-traumatic foot amputations are performed in diabetic patients. It is known that different mechanisms such as neuropathic degeneration (autonomic, motor, sensory), vasculopathy (micro and macroangiopathy), poorly controlled infection, and poor wound healing due to impaired collagen production are together in the etiopathogenesis of DA. In addition, opsonization and phagocytosis processes are reduced in diabetic patients. The decrease in chemotaxis and proliferation of cells responsible for inflammation and especially macrophages that stimulate wound healing by secreting various growth factors is one of the most important factors that delay wound healing. The characteristic feature in a diabetic foot case is a prolonged acute phase reaction. The first step in managing diabetic foot wounds is the evaluation, grading, and classification of the ulcer. There is no commonly agreed classification to be used in diabetic feet. Wagner-Meggit classification, San Antonio classification, University of Texas classification, PEDIS staging are a few of them. Each diabetic foot council uses its own appropriate classification. DA classification is an important guide in deciding on the treatment method and proceeding to amputation. Acute phase reactants such as C-reactive protein (CRP), white blood cell (WBC), neutrophil count, and sedimentation rate (ESR) are widely used as laboratory markers of progressing to amputation in DA, but these are insufficient to reflect the severity of DA disease. In addition, since no systemic effects can be seen in non-infected DA ulcers, an increase in acute-phase reactants may not be detected. For these reasons, new marker studies are needed to predict the prognosis of diabetic feet and determine the severity of the disease. Based on this need, investigators planned to examine the gremlin-1 level in DA foot cases in this study. Gremlin-1 is an extracellular antagonist of bone morphogenetic proteins (BMP) and works by directly neutralizing its ligands and inhibiting BMP signaling. BMP, a subgroup of TGF-B (transforming growth factor), an important pro-fibrinogenic cytokine, is known to have an anti-fibrinogenic role in various organs. BMP and its antagonist gremlin are developmental genes that regulate morphogenesis, and their role in embryogenesis has been clearly demonstrated in limb development, neural crest differentiation, and metanephric kidney organogenesis. Gremlin is silenced in adult tissues, but its induction in injured tissues has been described. Gremlin-1 expression has been shown to increase in pulmonary fibrosis, diabetic nephropathy, fibrotic liver diseases, and various malignancies. These findings indicate that Gremlin-1 plays a role in organ fibrosis. In addition, gremlin-1 plays a role in angiogenesis by binding to vascular endothelial factor receptor-2 (VEGFR-2) in endothelial cells. It is obvious that there is increased inflammation and accompanying fibrosis and angiogenesis during the healing process of DA wounds. Therefore, investigators aimed to examine the relationship between gremlin-1 levels and Wagner classification in DA cases and to test its usability as a biomarker in the progression to amputation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosed with DM
* Who either had diabetic foot ulcers or were at high risk for diabetic foot

Exclusion Criteria:

* Patients with autoimmune diseases
* Malignant conditions
* A history of prior amputation
* Those on hemodialysis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic foot who apply to the endocrinology outpatient clinic and are evaluated by the diabetic foot council.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
The increase in Wagner stage and the change in Gremlin-1 levels will be monitored and whether Gremlin-1 levels are a prognostic marker for predicting amputation in diabetic patients will be examined. | From enrollment to the end of physical exam and blood analysis at 10 months
  The Gremlin-1 levels of the patients included in the study will be evaluated between the groups according to their Wagner stage, and the statistical correlation between Wagner stage and Gremlin-1 will be investigated.
  Gremlin-1 levels will also be compared between amputee and non-amputee patients. It will be evaluated whether Gremlin-1 levels can be used as a prognostic marker in predicting amputation in diabetic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years after the publication of results

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT06753604/Prot_SAP_ICF_000.pdf